CLINICAL TRIAL: NCT04289116
Title: Enhancing Sexual Safety: Couples' Communication and HIV Testing Among YMSM
Acronym: WeTestATN156
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Hunter College of City University of New York (Other); Oregon Health and Science University (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Sylvie Naar, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ATN 156
Record Dates: First submitted 2020-02-14; First posted 2020-02-28 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: HIV/AIDS; HIV Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Intervention Model Description: At baseline participants will be randomized to one of two conditions: Condition 1: MI-CST + observation of ACT videos + CHTC, and Condition 2: Individual HIV Testing (IHTC) as usual. Youth have the choice of attending the baseline visit alone or with their partner and have the option to bring their partner in later after completing the baseline alone. Youth in this CET will complete follow-up assessments at 1, 3, and 6 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- We Test - Index Participants (Experimental): Each participant will receive MI-CST + observation of ACT videos + CHTC. Youth have the choice of attending the baseline visit alone or with their partner and have the option to bring their partner in later after completing the baseline alone.
  Interventions: Behavioral: We Test
- Individual HIV Testing and Counseling - Index Participants (Active Comparator): Individual HIV Testing and Counseling (IHTC). Youth have the choice of attending the baseline visit alone or with their partner and have the option to bring their partner in later after completing the baseline alone.
  Interventions: Behavioral: IHTC
- Individual Counseling and Testing - Partner Participants (Active Comparator): Referred partner who participates in Individual HIV Testing and Counseling with their partner.
  Interventions: Behavioral: IHTC

INTERVENTIONS:
Behavioral: We Test — This design tests the added benefits of adjunct intervention components delivered prior to receipt of CHTC-Assertive Communication Training (ACT) videos viewed by the couple separately and individually delivered Motivational Interviewing-based Communication Skills Training (MI-CST). These target the development of communication skills necessary to participate fully in HIV prevention and sexual safety discussions inherent to CHTC.
  Arms: We Test - Index Participants
Behavioral: IHTC — Individual HIV Testing and Counseling
  Arms: Individual Counseling and Testing - Partner Participants; Individual HIV Testing and Counseling - Index Participants

SUMMARY:
The purpose of this study is to compare different ways to deliver the couples HIV Testing and Counseling (CHTC) intervention that is suited for adolescents and young adults.

DETAILED DESCRIPTION:
Investigators will conduct a comparative effectiveness trial (CET) of CHTC for adolescent-age (15-24 years) same-sex male couples. This design tests the added benefits of adjunct intervention components delivered prior to receipt of CHTC-Assertive Communication Training (ACT) videos viewed by the individual or couple together and individually delivered Motivational Interviewing-based Communication Skills Training (MI-CST). These target the development of communication skills necessary to participate fully in HIV prevention and sexual safety discussions inherent to CHTC. Youth will be randomized to receive one of two conditions: Condition 1: watch videos on ACT, participate in Communication Skills Training (MI-CST), and complete an individual HIV test, or if participating as a couple will receive CHTC, and Condition 2: Individual HIV Testing (IHTC) as usual. Youth have the choice of attending the baseline visit alone or with their partner and have the option to bring their partner in later after completing the baseline alone. Youth in this CET will complete follow-up assessments at 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* At least one partner must be HIV-negative or status unknown
* THE INDEX PARTNER must be 15-24 years old
* YMSM under age 18 MUST HAVE AN AGE CONCORDANT PARTNER TO PARTICIPATE IN THIS STUDY, I.E., MINORS may only participate in the study with a partner within 2 years of age OF THE MINOR SUBJECT'S AGE. THE AGE CONCORDANT PARTNER MUST BE AT LEAST FIFTEEN YEARS OLD.
* INDEX PARTNER MUST BE SEXUALLY ACTIVE (ANY ACTIVITY THAT COULD LEAD TO ORGASM)
* CURRENTLY SEEING SOMEONE, DATING, EXPERIMENTING WITH RELATIONSHIPS OR IN A RELATIONSHIP
* HAVE HAD SEX, HOOKED UP WITH OR MADE OUT WITH THAT PERSON
* Both partners must be able to communicate in English.
* LIVE IN OR NEAR NEW YORK CITY OR DETROIT OR SAN DIEGO
* GENDER IDENTITY AS MALE OR nonbinary, GENDERQUEER, agender OR GENDER NONCOMFORMING

Exclusion Criteria:

* Unstable, serious psychiatric symptoms
* Current suicidal/homicidal ideation
* Current or prior Intimate Partner Violence (IPV) on the part of either relationship partner
* IF EITHER PARTICIPATING PARTNER FELT PRESSURED OR COERCED TO PARTICIPATE IN THE STUDY OR FELT ANYONE MADE THEM FEEL THEY HAD TO PARTICIPATE IN THEY STUDY WHEN THEY DID NOT WANT TO.

Ages: 15 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Identifies as male, nonbinary, genderqueer or gender nonconforming.
Enrollment: 71 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyrel Starks, PhD, Study Chair — City University of New York; Sarah W Feldstein Ewing, PhD, Study Chair — University of Rhode Island
Locations (2):
- United States (2):
  - Wayne State University, Detroit, Michigan
  - The City University of New York, New York, New York

IPD SHARING:
Plan to Share IPD: No
Currently, there is no plan to share the study data at this time; however, the study team is currently in the process of developing a plan to share data, while protecting the privacy and confidentiality of participants.

RESULTS

PARTICIPANT FLOW:
Groups:
- We Test - Index Participants: Each individual who attended We Test received MI-CST + observation of ACT videos + CHTC. Youth have the choice of attending the baseline visit alone or with their partner and have the option to bring their partner in later after completing the baseline alone.
  We Test: This design tests the added benefits of adjunct intervention components delivered prior to receipt of CHTC-Assertive Communication Training (ACT) videos viewed by the couple separately and individually delivered Motivational Interviewing-based Communication Skills Training (MI-CST). These target the development of communication skills necessary to participate fully in HIV prevention and sexual safety discussions inherent to CHTC.
- Individual HIV Testing and Counseling - Index Participants: Individual HIV Testing and Counseling (IHTC). Youth have the choice of attending the baseline visit alone or with their partner and have the option to bring their partner in later after completing the baseline alone. This includes 1 index partner who completed the intervention with their partner.
  IHTC: Individual HIV Testing and Counseling
- Individual Counseling and Testing - Partner Participants: Youth have the choice of attending the baseline visit alone or with their partner and have the option to bring their partner in later after completing the baseline alone. Only 1 couple chose this option. This couple attended the intervention together and received individual HIV testing and counseling.
Period: Overall Study
Arm/Group | We Test - Index Participants | Individual HIV Testing and Counseling - Index Participants | Individual Counseling and Testing - Partner Participants
Started | 33 | 37 | 1
Completed | 33 | 37 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | We Test - Index Participants | Individual HIV Testing and Counseling - Index Participants | Individual Counseling and Testing - Partner Participants | Total
Number analyzed (Participants) | 33 | 37 | 1 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.91 (1.86) | 22.38 (1.77) | 24.00 | 22.18 (1.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 33 | 37 | 1 | 71
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 4 | 11 | 0 | 15
  Latino | 13 | 9 | 0 | 22
  White | 13 | 12 | 1 | 26
  Other | 3 | 5 | 0 | 8
Sexual Identity [Count of Participants; unit: Participants]
  Gay | 23 | 25 | 1 | 49
  Other/Queer | 10 | 12 | 0 | 22
Gender Identity [Count of Participants; unit: Participants]
  Cisgender Male | 26 | 30 | 1 | 57
  Transgender, gender nonconforming, or assigned male at birth | 7 | 7 | 0 | 14
Employment [Count of Participants; unit: Participants]
  Yes | 22 | 26 | 1 | 49
  No | 11 | 11 | 0 | 22
Health Insurance [Count of Participants; unit: Participants]
  No | 5 | 5 | 0 | 10
  Yes, my own | 14 | 16 | 0 | 30
  Yes, my guardian | 14 | 16 | 1 | 31
Current PrEP Use [Count of Participants; unit: Participants]
  No | 21 | 25 | 1 | 47
  Yes | 12 | 12 | 0 | 24
Main Partner Age [Mean (Standard Deviation); unit: Years] | 25.45 (7.89) | 26.11 (6.59) | 24.00 (0.00) | 25.77 (7.14)
Relationship Length (in months) [Mean (Standard Deviation); unit: Months] | 19.21 (25.03) | 21.14 (26.56) | 2.00 (0.00) | 19.97 (25.59)

OUTCOME MEASURES:

1. Primary Outcome: HIV Transmission Risk Behavior
Description: Self-reported Condomless anal sex with a casual partner
Time Frame: baseline, month 3, month 6
Population: Intent to treat population. Analysis only includes participants who participated in the We Test - Index arm and Individual HIV Testing and Counseling - Index arm on their own.
Measure: Count of Participants; unit: Participants
Groups:
- We Test - Index Participants: Each participant or couple will receive MI-CST + observation of ACT videos + CHTC. Youth have the choice of attending the baseline visit alone or with their partner and have the option to bring their partner in later after completing the baseline alone.
  We Test: This design tests the added benefits of adjunct intervention components delivered prior to receipt of CHTC-Assertive Communication Training (ACT) videos viewed by the couple separately and individually delivered Motivational Interviewing-based Communication Skills Training (MI-CST). These target the development of communication skills necessary to participate fully in HIV prevention and sexual safety discussions inherent to CHTC.
Arm/Group | We Test - Index Participants | Individual HIV Testing and Counseling - Index Participants | Individual Counseling and Testing - Partner Participants
Number analyzed (Participants) | 33 | 37 | 1
Participants
  Baseline | 9 | 11 | 0
  3 month: number analyzed (Participants) | 33 | 37 | 0
  3 month | 4 | 8 | 0
  6 month | 4 | 6 | 0
Statistical Analysis 1: Comparison: We Test - Index Participants vs Individual HIV Testing and Counseling - Index Participants; Analysis only includes participants who participated in the We Test - Index arm and Individual HIV Testing and Counseling - Index arm on their own; Test type: Superiority; p = 0.20, Negative Binomial Regression; Chi Square = 1.36
Statistical Analysis 2: Comparison: We Test - Index Participants vs Individual HIV Testing and Counseling - Index Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.58, Negative Binomial Regression; Chi Square = 0.03

2. Secondary Outcome: Communication Skills
Description: Interpersonal Communication Competence Scale, higher scores are associated with better communication skills, range 0 - 150.
Time Frame: baseline, month 3, month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | We Test - Index Participants | Individual HIV Testing and Counseling - Index Participants | Individual Counseling and Testing - Partner Participants
Number analyzed (Participants) | 33 | 37 | 1
Units on a scale
  Baseline | 123 (11.01) | 121.19 (12.78) | 129.00
  3 month: number analyzed (Participants) | 33 | 37 | 0
  3 month | 125.04 (10.04) | 119.04 (12.97) |
  6 month | 125.27 (12.81) | 117.68 (11.30) | 129.00
Statistical Analysis 1: Comparison: We Test - Index Participants vs Individual HIV Testing and Counseling - Index Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.08, t-test, 2 sided; Mean Difference (Final Values) = -1.82
Statistical Analysis 2: Comparison: We Test - Index Participants vs Individual HIV Testing and Counseling - Index Participants; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.02, t-test, 2 sided; Mean Difference (Final Values) = -2.5

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | We Test - Index Participants | Individual HIV Testing and Counseling - Index Participants | Individual Counseling and Testing - Partner Participants
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/37 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/37 | 0/1
Other Adverse Events (participants affected / at risk) | 0/33 | 0/37 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT04289116/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT04289116/SAP_001.pdf
  • Informed Consent Form (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT04289116/ICF_002.pdf